CLINICAL TRIAL: NCT04711291
Title: Efficacy of Envarsus XR and Digital Health Technology in Reducing Tacrolimus Fluctuation and Frequency of Dose Changes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left organization and study not adopted by any other staff.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020P001109
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Medication Adherence; Renal Transplant
Keywords: QR code technology; Envarsus-XR; Tacrolimus trough level; Digital health technology
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: BIDMC kidney transplant patients currently taking immediate release tacrolimus (IR-Tac) will be screened for enrollment into the trial. Eligible patients will be randomized to one of three treatment arms in a 1:1:1 fashion. We aim to randomize seventy-five (75) patients into one of three treatment arms (1:1:1) as described.
  Arm 1: Remain on tacrolimus immediate release (IR-Tac) prescribed doses every 12 hours; Arm 2: Convert to tacrolimus extended release (Envarsus XR) prescribed dose every 24 hours; OR Arm 3: Convert to tacrolimus extended release (Envarsus XR) prescribed dose every 24 hours used in combination with the smart phone application, TransMedAxTM.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Remain on IR-Tac prescribed doses every 12 hours (No Intervention): Patient will remain in Tacrolimus IR-Tac Arm and will complete medication adherence questionnaire monthly. They will not receive any notifications from TransMedAx application. Research staff and PI will collect their Tacrolimus Trough levels and change in tacrolimus dose levels during their routine follow up.
- Convert to Envarsus XR once daily (Active Comparator): Subjects randomized to this arm will switch from IR-Tac to Envarsus XR and will complete medication adherence questionnaire. However, patients in this group will not receive any notifications from TransMedAx application. Research staff and PI will collect their Tacrolimus trough levels and change in tacrolimus dose during their follow up.
  Interventions: Drug: Convert to Envarsus XR once daily
- Convert to Envarsus XR once daily combined with TransMedAx app use (Experimental): Subjects randomized to this arm will switch from IR-Tac to Envarsus XR, will receive notification by scanning a QR code through TransMedAx application and will complete medication adherence questionnaire. Research staff and PI will collect their Tacrolimus trough levels and change in tacrolimus dose during their follow up.
  Interventions: Combination Product: Conversion to Envarsus-XR and use of smart phone app, TransMedAx

INTERVENTIONS:
Combination Product: Conversion to Envarsus-XR and use of smart phone app, TransMedAx — Convert to tacrolimus extended release (Envarsus XR) prescribed dose every 24 hours used in combination with the smart phone application, TransMedAx.
  Patients in this arm will be trained to use the app along with conversion to Envarsus-XR. Once patient scan the code on medicine bottle and the app will remind them about the time and dose of the medication in their native language.
  Arms: Convert to Envarsus XR once daily combined with TransMedAx app use
Drug: Convert to Envarsus XR once daily — Convert from tacrolimus immediate release to tacrolimus extended release (Envarsus XR) prescribed dose every 24 hours
  Arms: Convert to Envarsus XR once daily

SUMMARY:
Tacrolimus is an immunosuppressive agent prescribed to prevent organ rejection in post transplant patients, in combination with other immunosuppressants. In post-kidney transplant patients, tacrolimus blood trough(peak) level must be monitored frequently, and dose adjustments must be made as necessary to keep trough level within a very narrow target range.

High tacrolimus intra-patient variability(IPV) can be a marker of medication non-adherence. The presence of medication non-adherence could be due to multiple factors e.g. Forgetfulness, misunderstanding or miscommunication due to language barrier etc. Our hypothesis is using QR code technology along with extended release Tacrolimus medication will reduce tacrolimus IPV fluctuation.

DETAILED DESCRIPTION:
Tacrolimus is a calcineurin-inhibitor immunosuppressant indicated for the prophylaxis of organ rejection in patients receiving allogeneic liver, kidney or heart transplants, in combination with other immunosuppressants. Envarsus XR (extended release tacrolimus) is a long acting form of tacrolimus that is prescribed as a single dose per day (every 24 hours) rather than immediate release tacrolimus (IR-Tac) which is prescribed as a two doses per day (every 12 hours).

In post-kidney transplant patients, tacrolimus blood trough level must be monitored frequently, and dose adjustments must be made as necessary to keep trough level within a very narrow therapeutic range. High intra-patient variability (IPV) has also been reported to promote donor-specific antibody development, increased graft rejection rates and poor long-term outcome after kidney transplantation. In addition to increased potential for poor graft outcomes, these fluctuations and frequent dose adjustments are confusing and burdensome for patients, add to costs via medication expenses and need for lab checks, and consume the limited resources of transplant centers.

Similarly, non-adherence with immunosuppression medications is common and also linked to poor graft outcomes in kidney transplant patients.

High tacrolimus IPV can be a marker of medication non-adherence. The presence of medication non-adherence could be due to multiple factors such as forgetfulness to take the medication or remembering the correct dose, misunderstanding or miscommunication due to language barrier or logistical issues. High tacrolimus IPV could also be due to difficulty in taking medication every 12 hours, variation in bioavailability of different generic tacrolimus formulations or drug interactions. Considering the IPV of Tacrolimus level, patients and their families often have difficulty managing medications, especially during frequent changes in medication doses. This problem is more prevalent for older patients, who are often on multiple medications and for whom side effects and drug-drug interactions may lead to more harm. Once daily tacrolimus has had mixed results in reducing tacrolimus IPV. Very few studies have been done till now to measure the IPV among patients who received twice daily IR-Tac and converted to once daily Envarsus-XR. These studies were able to show significant reduction in IPV among patients who had high IPV prior to conversion. It is also noteworthy as compared to Astragraf, Envarsus XR has a more favorable pharmacokinetic profile. Envarsus XR uses Melt Dose technology to increase bioavailability and allow a more controlled release of the drug. This results in less fluctuation between maximum ("peak") exposure and trough. From a clinical perspective, Envarsus is noninferior in terms of efficacy (composite endpoint, including kidney transplant graft loss, death, biopsy-proven acute rejection and loss to follow-up) when compared to IR-Tac with a similar safety profile.

Digital health technologies have not been studied in regards to tacrolimus IPV but have shown promising results in improving medication adherence, including in kidney transplant population. TransMedAxTM application; a proposed digital health platform that will be developed to be used in this study. It will utilize dynamic QR code based technology customized to each individual patient, to improve medication adherence. It is especially geared towards patient populations who have frequent changes in medication dosages and have limited English language proficiency. A brief description of TransMedAxTM workflow is as follows:

* Patients will be asked to bring their medication bottle/pill box to the clinic. A QR code unique to the patient will be printed from TransMedAxTM website and attached to medication bottle. TransMedAxTM app will be downloaded on patient's phone.
* Research staff will input tacrolimus medication and dose into the patient's TransMedAxTM application account. The TransMedAxTM verbal instructions will be automatically translated into the patient's preferred language (English, Spanish, Haitian/Creole, or Mandarin).

When this QR code is scanned by the patient using their smartphone camera, it will provide verbal instructions on Tacrolimus dosage and also display the time of the dose on patient's phone. The TransMedAxTM application installed on patient's phone home screen will allow patient to access this information at one-tap and send reminders when the tacrolimus is due. This application will also be used to monitor patient adherence using brief questionnaire.

Many patients and clinicians hope technology will help improve safety, but technology may increase errors if not properly implemented.

Our project will specifically focus on transplant patients in their home/outpatient setting, and addresses language barrier for communication, coordination, and information for these patients. Our focus is on improving patient self-management of tacrolimus medication and informed partnership with clinicians to improve safety.

If successful, our work will have the following impact:

* Provide patients/families, and providers with a readily available tool to manage Tacrolimus doses.
* Improve adherence to the immunosuppressive therapy at appropriate doses prescribed by physician on timely manner.
* This measures will reduce the rate of acute rejection, graft loss and drug side effects and hence the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. BIDMC adult kidney transplant recipient more than 2 years post transplant
2. On tacrolimus IR regimen
3. Estimated glomerular filtration rate (eGFR) >45
4. Tacrolimus dose adjustments 2 or more times in past 12 months
5. Own and able to use a smart phone.
6. Able to consent

Exclusion Criteria:

1. Prisoners
2. Patients with primary language other than English, Spanish, Haitian/Creole, Mandarin
3. Patients who can't swallow whole tablets or capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of tacrolimus dose changes in 12 month period. | 1 year follow up
  How frequent was the dose changes in 12 month follow up post transplant, excluding changes made due to change in therapeutic target.

SECONDARY OUTCOMES:
Change in number of tacrolimus dose adjustments in follow up period compared to 12 months prior to enrolment, excluding changes made due to change in therapeutic target | 12 months
  We will note the change in number of Tacrolimus dose adjustments in follow up period and compared the dose changes 12 months prior to enrollment. We will exclude the changes made due to change in therapeutic target.
Self-reported adherence via monthly questionnaire. | 12 months
  We will monitor the patient compliance with self medications among arms and note frequency of non adherence.
• Variability in tacrolimus trough levels, as checked on routine labs as part of standard care | 12 months
  We will monitor the fluctuations in Tacrolimus Trough levels among patients randomized to different arms and compared their variability with the one in Arm 3

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Agrawal, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Martha Pavlakis, MD, Study Director — Beth Israel Deaconess Medical Center; Amtul Aala, MD, Study Chair — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borra LC, Roodnat JI, Kal JA, Mathot RA, Weimar W, van Gelder T. High within-patient variability in the clearance of tacrolimus is a risk factor for poor long-term outcome after kidney transplantation. Nephrol Dial Transplant. 2010 Aug;25(8):2757-63. doi: 10.1093/ndt/gfq096. Epub 2010 Feb 26. PMID 20190242
- [Background] Kahan BD, Welsh M, Urbauer DL, Mosheim MB, Beusterien KM, Wood MR, Schoenberg LP, Dicesare J, Katz SM, VAN Buren CT. Low intraindividual variability of cyclosporin A exposure reduces chronic rejection incidence and health care costs. J Am Soc Nephrol. 2000 Jun;11(6):1122-1131. doi: 10.1681/ASN.V1161122. PMID 10820177
- [Background] Sapir-Pichhadze R, Wang Y, Famure O, Li Y, Kim SJ. Time-dependent variability in tacrolimus trough blood levels is a risk factor for late kidney transplant failure. Kidney Int. 2014 Jun;85(6):1404-11. doi: 10.1038/ki.2013.465. Epub 2013 Dec 11. PMID 24336032
- [Background] Shen CL, Yang AH, Lien TJ, Tarng DC, Yang CY. Tacrolimus Blood Level Fluctuation Predisposes to Coexisting BK Virus Nephropathy and Acute Allograft Rejection. Sci Rep. 2017 May 16;7(1):1986. doi: 10.1038/s41598-017-02140-1. PMID 28512328
- [Background] Shuker N, Cadogan M, van Gelder T, Roodnat JI, Kho MM, Weimar W, Hesselink DA. Conversion from twice-daily to once-daily tacrolimus does not reduce intrapatient variability in tacrolimus exposure. Ther Drug Monit. 2015 Apr;37(2):262-9. doi: 10.1097/FTD.0000000000000136. PMID 25265255
- [Background] Rostaing L, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT Jr, Budde K; Envarsus Study Group. Novel Once-Daily Extended-Release Tacrolimus Versus Twice-Daily Tacrolimus in De Novo Kidney Transplant Recipients: Two-Year Results of Phase 3, Double-Blind, Randomized Trial. Am J Kidney Dis. 2016 Apr;67(4):648-59. doi: 10.1053/j.ajkd.2015.10.024. Epub 2015 Dec 22. PMID 26717860
- [Background] Foster BJ, Pai ALH, Zelikovsky N, Amaral S, Bell L, Dharnidharka VR, Hebert D, Holly C, Knauper B, Matsell D, Phan V, Rogers R, Smith JM, Zhao H, Furth SL. A Randomized Trial of a Multicomponent Intervention to Promote Medication Adherence: The Teen Adherence in Kidney Transplant Effectiveness of Intervention Trial (TAKE-IT). Am J Kidney Dis. 2018 Jul;72(1):30-41. doi: 10.1053/j.ajkd.2017.12.012. Epub 2018 Mar 27. PMID 29602631
- [Background] Riley-Lawless K. Family-identified barriers to medication reconciliation. J Spec Pediatr Nurs. 2009 Apr;14(2):94-101. doi: 10.1111/j.1744-6155.2009.00182.x. PMID 19356203
- [Background] Manias E, Hughes C. Challenges of managing medications for older people at transition points of care. Res Social Adm Pharm. 2015 May-Jun;11(3):442-7. doi: 10.1016/j.sapharm.2014.10.001. Epub 2014 Oct 13. PMID 25455760
- [Background] Quintana Y, Fahy D, Crotty B, Jain R, Kaldany E, Gorenberg M, Lipsitz L, Engorn D, Rodriguez J, Orfanos A, Bajracharya A, Henao J, Adra M, Skerry D, Slack WV, Safran C. InfoSAGE: Supporting Elders and Families through Online Family Networks. AMIA Annu Symp Proc. 2018 Dec 5;2018:932-941. eCollection 2018. PMID 30815136
- [Background] Quintana Y, Crotty B, Fahy D, Lipsitz L, Davis RB, Safran C. Information sharing across generations and environments (InfoSAGE): study design and methodology protocol. BMC Med Inform Decis Mak. 2018 Nov 20;18(1):105. doi: 10.1186/s12911-018-0697-4. PMID 30458840
- [Background] Quintana Y, Gonzalez Martorell EA, Fahy D, Safran C. A Systematic Review on Promoting Adherence to Antiretroviral Therapy in HIV-infected Patients Using Mobile Phone Technology. Appl Clin Inform. 2018 Apr;9(2):450-466. doi: 10.1055/s-0038-1660516. Epub 2018 Jun 20. PMID 29925099
- [Background] Wolfstadt JI, Gurwitz JH, Field TS, Lee M, Kalkar S, Wu W, Rochon PA. The effect of computerized physician order entry with clinical decision support on the rates of adverse drug events: a systematic review. J Gen Intern Med. 2008 Apr;23(4):451-8. doi: 10.1007/s11606-008-0504-5. PMID 18373144
- [Background] Langone A, Steinberg SM, Gedaly R, Chan LK, Shah T, Sethi KD, Nigro V, Morgan JC; STRATO Investigators. Switching STudy of Kidney TRansplant PAtients with Tremor to LCP-TacrO (STRATO): an open-label, multicenter, prospective phase 3b study. Clin Transplant. 2015 Sep;29(9):796-805. doi: 10.1111/ctr.12581. Epub 2015 Aug 6. PMID 26113208